CLINICAL TRIAL: NCT05217394
Title: Evaluating the Effectiveness of the Occupational Therapy Handwriting Intervention Guideline on Handwriting Skills for Children: A Protocol for Clustered-Randomised Control Trial
Brief Title: Effectiveness of the Occupational Therapy Handwriting Intervention Guideline on Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: Ministry of Education, Malaysia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FRGS/1/2020/SSI0/UKM/03/2
Record Dates: First submitted 2022-01-09; First posted 2022-02-01 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Difficulty Writing
Keywords: handwriting; intervention; effectiveness; children; study protocol; clustered randomized controlled trial

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OTHIG (Experimental): Occupational Therapy Handwriting Intervention Guideline - this is the experimental guideline to be tested in this study.
  Section C: Intervention for Handwriting Readiness Skills
  * Handwriting development
  * Pre-writing skills
  * Gross motor skills activities
  * Fine motor skills activities
  * Motor visual skills activities Section D: Intervention for Handwriting Skills
  * Handwriting tools
  * Pencil grasp
  * Posture and position
  * Hand dominance
  * Writing capitals, lowercase, and numbers
  * Handwriting speed Section E: Handwriting Intervention Module
  * Session 1: Development of Handwriting Skills Activities
  * Session 2: Pre-writing Skills Activities
  * Session 3: Gross and Fine Motor Skills Activities
  * Session 4: Writing Capital Letters
  * Session 5: Writing Lowercase Letters
  * Session 6: Writing Numbers
  Interventions: Other: OTHIG
- NOTi (No Intervention): Natural Occupational Therapy Intervention - this means, the participants in this group are not exposed to the OTHIG. They receive natural OT intervention without exposure to the OTHIG.
  The natural OT intervention includes:
  Gross motor skills, fine motor skills, pre-writing skills, basic handwriting tasks such as copying, tracing, imitating and colouring.
  It will follow the occupational therapist intervention set up by the respected therapist in charge. The OT in charge had qualifications from the local university in Malaysia.
  The natural OT intervention includes:
  Gross motor skills, fine motor skills, pre-writing skills, basic handwriting tasks such as copying, tracing, imitating and colouring.
  It will follow the occupational therapist intervention set up by the respected therapist in charge. The OT in charge had qualifications from the local university in Malaysia.

INTERVENTIONS:
Other: OTHIG — Occupational Therapy Handwriting Intervention Guideline
  Arms: OTHIG

SUMMARY:
This study aims to evaluate the effectiveness of the Occupational Therapy Handwriting Interventions Guidelines (OTHIG) in enhancing handwriting performance among children.

Method:

Forty-two children recruited from private centers with occupational therapy indications and with handwriting issues, aged five to nine years, will be assigned to the experimental and control groups.

Participants will receive a total of 10-week sessions, including training, intervention, and outcome measures.

The experimental group will receive the developed OTHIG during handwriting skills intervention. Meanwhile, the control group will receive conventional interventions which not exposed to the OTHIG.

This study is expected to provide evidence for the effectiveness of using the developed OTHIG to OTs in delivering their services, targeting children struggling with handwriting skills.

DETAILED DESCRIPTION:
The study is a Cluster Randomised Controlled Trial (C-RCT) that systematically clusters the centers into the treatment and control groups.

A total of 10 centers will be involved in this study.

The clustering of all ten centers will allocate randomly into the treatment and control groups based on submitting the consent letter to the researcher and after an assessment of TPT and TVPS-4 are conducted.

Ten early interventions have similar characteristics such as (1) hiring graduated occupational therapists from recognized universities in Malaysia, (2) having occupational therapists working daily at the centre, (3) having children aged five to nine years who receive OTs intervention.

This randomization will be allocated based on the list of the centers that give an early submission of a signed consent form. The randomization will be carried out with a mechanism that neither the researcher nor children or center owners will know which group of intervention they will be assigned.

ELIGIBILITY:
Inclusion Criteria:

* age between five and nine years
* engaged in OTs intervention either in an individual or group session.

Exclusion Criteria:

* refuse to participate in the study
* fail to comply with the whole intervention process during the study
* present severe sensory problems
* present poor behavior during intervention

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
The Print Tool | 2 weeks
  Handwriting assessment

SECONDARY OUTCOMES:
Test of Visual Perceptual Skills-4 | 2 weeks
  Visual perceptual skills assessment

CONTACTS AND LOCATIONS:
Overall Officials: Masne Kadar, Study Director — Faculty of Health Sciences, UKM
Locations (4):
- Malaysia (4):
  - Kiddie Care Centre, Jitra, Kedah
  - Ryan Special Needs Rehabilitation Centre, Putrajaya, PU
  - Excel Qhalif Playgroup Centre, Bangi, Selangor
  - Kizzu Kids Centre, Shah Alam, Selangor

IPD SHARING:
Plan to Share IPD: Yes
All data collected will be shared among researchers
Supporting Information: Study Protocol
Time Frame: October 2021 until September 2022
Access Criteria: Study protocol will be shared with all researchers

DOCUMENTS (2):
  • Study Protocol (2022-09-25): https://cdn.clinicaltrials.gov/large-docs/94/NCT05217394/Prot_002.pdf
  • Informed Consent Form (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT05217394/ICF_001.pdf